CLINICAL TRIAL: NCT02986269
Title: The Value of Pressure Support on Ventilation Inhomogeneity and Lung Function in Patients Under Spontaneous Breathing (SB)Across Laryngeal Mask Airway
Brief Title: PSV on Ventilation Inhomogeneity and Lung Function in Patients Under SB Across LMA
Acronym: VINHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walid HABRE (Other)
Responsible Party: Sponsor-Investigator, Walid HABRE, Anesthesiology, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: VINHO
Record Dates: First submitted 2016-11-25; First posted 2016-12-08 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Respiratory Function Tests; Anesthesia, General; Patient Positioning; Ventilation
Keywords: Respiratory Function; Patient Positioning; anesthesia
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SB (Experimental): Patient is scheduled for elective conisation or hysteroscopy under general anesthesia. The ventilation mode for this group is spontaneous breathing(SB) without pressure support ventilation (PSV) under laryngeal mask airway (LMA).
  General anesthesia across LMA under SB without PSV
  Interventions: Procedure: general anesthesia across LMA; Procedure: Spontaneous breathing(SB)
- Group PSV (Active Comparator): General anesthesia across LMA under SB with PSV Patient is scheduled for elective conisation or hysteroscopy under general anesthesia. The ventilation mode for this group is SB with PSV under LMA.
  Interventions: Procedure: general anesthesia across LMA; Procedure: Spontaneous breathing(SB); Procedure: Pressure Support Ventilation

INTERVENTIONS:
Procedure: general anesthesia across LMA — general anesthesia across LMA
Procedure: Spontaneous breathing(SB) — general anesthesia across LMA under SB without PSV
Procedure: Pressure Support Ventilation — general anesthesia across LMA under SB with PSV
  Arms: Group PSV

SUMMARY:
General anesthesia has been demonstrated to have a negative impact on lung function. Both surgery and patient position influence the perioperative lung function. Laryngeal mask airway (LMA) has been proved to be safe and efficient to maintain the airways patent during general anesthesia. Pressure support ventilation (PSV) with LMA is routinely used in clinical practice. The aim of the present trial is to characterize perioperative changes in lung volume, ventilation inhomogeneity and respiratory mechanics in patients in the lithotomy position and spontaneously breathing through LMA with and without PSV.

DETAILED DESCRIPTION:
This study is a randomized controlled trial. Participants for this study will be recruited from the Gynecological department of the University Hospitals of Geneva, scheduled for gynecological procedures in the lithotomy position under general anesthesia. A total of 40 patients will be enrolled and randomly assigned into 2 groups: Group SB (spontaneously breathing without PSV) and Group PSV (spontaneously breathing with PSV). Measurements of end-expiratory lung volume (EELV) and ventilation inhomogeneity will be performed in all patients with a nitrogen multiple breath washout method, before and 1 hour after surgery. Similarly, airway resistance (Rrs) and reactance (Xrs) will be measured at the same time by using the Forced Oscillation Technique.

The primary endpoint: Perioperative changes in ventilation inhomogeneity (LCI) and respiratory mechanics (Rrs and Xrs) of patients, positioned in lithotomy and undergoing general anesthesia while breathing spontaneously through LMA with or without PSV.

The secondary endpoints: Presence of respiratory complications, oxygen need in the recovery room, length of stay in the recovery room and in the hospital. Correlation between duration of positioning and surgery with lung function and volume measurements.

Relevance: There are no studies that addressed the value of pressure support ventilation to overcome the potential changes in lung function following spontaneous ventilation across a LMA in the lithotomy position.

ELIGIBILITY:
Inclusion Criteria:

- American Society of Anesthesiologists physical status (ASA) Ⅰ and Ⅱ grade, adult female patients, aged between 18 and 50 years scheduled for elective gynecological surgery in the lithotomy position.

Exclusion Criteria:

1. Age<18 years and >50 years old
2. ASA score of III-V
3. Patients with a potentially difficult airway (cervical spine disease, Mallampati classification III or IV or mouth opening of <2.5 cm)
4. Risk of regurgitation/aspiration(previous upper gastrointestinal tract surgery, known or symptomatic hiatus hernia, oesophageal reflux, peptic ulceration or not fasted)
5. Respiratory diseases(bronchial asthma requiring therapy)
6. Patient refusal
7. Malignant hyperthermia history
8. Sore throat within 10 days
9. Body mass index (BMI) >30 kg/m2
10. Cardiac disease associated with dyspnea more than New York Heart Association II
11. Severe psychiatric disorder.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Perioperative changes in ventilation inhomogeneity (LCI) | Through study completion, an average of 12 hours
  LCI will be derived from the nitrogen multiple breath washout technique that will be applied before and after general anesthesia for gynecology in the lithotomy position with patients breathing spontaneously through a LMA with and without pressure support.

SECONDARY OUTCOMES:
Alterations in end expiratory lung volume in ml/kg (EELV) | Through study completion, an average of 12 hours
  EELV will be measured from the nitrogen multiple breath washout technique that will be applied before and after general anesthesia for gynecology in the lithotomy position with patients breathing spontaneously through a LMA with and without pressure support.
Changes in respiratory system compliance (Crs) | Through study completion, an average of 12 hours
  Crs will be measured by the forced oscillation technique
Changes in airway resistance (Raw) | Through study completion, an average of 12 hours
  Raw will be measured by the forced oscillation technique
Perioperative respiratory complications | Through study completion, an average of 12 hours
  any respiratory complications (apnoea/ bradypnoea, bronchospasm, laryngospasm, oxygen desaturation <90%/ hypoxemia, hypoventilation/ atelectasis, pulmonary embolism, cough and /or airway obstruction

CONTACTS AND LOCATIONS:
Overall Officials: Walid HABRE, MD,PhD, Principal Investigator — University Hospitals of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tiefenthaler W, Pehboeck D, Hammerle E, Kavakebi P, Benzer A. Lung function after total intravenous anaesthesia or balanced anaesthesia with sevoflurane. Br J Anaesth. 2011 Feb;106(2):272-6. doi: 10.1093/bja/aeq321. Epub 2010 Nov 9. PMID 21062790
- [Result] Daley MD, Norman PH, Colmenares ME, Sandler AN. Hypoxaemia in adults in the post-anaesthesia care unit. Can J Anaesth. 1991 Sep;38(6):740-6. doi: 10.1007/BF03008452. PMID 1914057
- [Result] von Ungern-Sternberg BS, Regli A, Schneider MC, Kunz F, Reber A. Effect of obesity and site of surgery on perioperative lung volumes. Br J Anaesth. 2004 Feb;92(2):202-7. doi: 10.1093/bja/aeh046. PMID 14722169
- [Result] Grocott HP. From the Journal archives: Airway closure and lung volumes in surgical positions. Can J Anaesth. 2014 Apr;61(4):383-6. doi: 10.1007/s12630-013-0098-1. Epub 2014 Jan 18. PMID 24442988
- [Result] Reber A, Bein T, Hogman M, Khan ZP, Nilsson S, Hedenstierna G. Lung aeration and pulmonary gas exchange during lumbar epidural anaesthesia and in the lithotomy position in elderly patients. Anaesthesia. 1998 Sep;53(9):854-61. doi: 10.1046/j.1365-2044.1998.00491.x. PMID 9849278
- [Result] Brain AI. The laryngeal mask--a new concept in airway management. Br J Anaesth. 1983 Aug;55(8):801-5. doi: 10.1093/bja/55.8.801. PMID 6349667
- [Result] Keller C, Brimacombe J. [Spontaneous versus controlled respiration with the laryngeal mask. A review]. Anaesthesist. 2001 Mar;50(3):187-91. doi: 10.1007/s001010050987. German. PMID 11315492
- [Result] Keller C, Sparr HJ, Brimacombe JR. Positive pressure ventilation with the laryngeal mask airway in non-paralysed patients: comparison of sevoflurane and propofol maintenance techniques. Br J Anaesth. 1998 Mar;80(3):332-6. doi: 10.1093/bja/80.3.332. PMID 9623433
- [Result] Radhika KS, Sripriya R, Ravishankar M, Hemanth Kumar VR, Jaya V, Parthasarathy S. Assessment of suitability of i-gel and laryngeal mask airway-supreme for controlled ventilation in anesthetized paralyzed patients: A prospective randomized trial. Anesth Essays Res. 2016 Jan-Apr;10(1):88-93. doi: 10.4103/0259-1162.167849. PMID 26957697
- [Result] Sharma R, Dua CK, Saxena KN. A randomised controlled study comparing the effects of laryngeal mask airway and endotracheal tube on early postoperative pulmonary functions. Singapore Med J. 2011 Dec;52(12):874-8. PMID 22159929
- [Result] Capdevila X, Jung B, Bernard N, Dadure C, Biboulet P, Jaber S. Effects of pressure support ventilation mode on emergence time and intra-operative ventilatory function: a randomized controlled trial. PLoS One. 2014 Dec 23;9(12):e115139. doi: 10.1371/journal.pone.0115139. eCollection 2014. PMID 25536515
- [Result] Keller C, Brimacombe J, Hoermann C, Loeckinger A, Kleinsasser A. Pressure support ventilation with the ProSeal laryngeal mask airway. A comparison of sevoflurane, isoflurane and propofol. Eur J Anaesthesiol. 2005 Aug;22(8):630-3. doi: 10.1017/s0265021505001055. PMID 16119601
- [Result] Chiumello D, Pelosi P, Calvi E, Bigatello LM, Gattinoni L. Different modes of assisted ventilation in patients with acute respiratory failure. Eur Respir J. 2002 Oct;20(4):925-33. doi: 10.1183/09031936.02.01552001. PMID 12412685
- [Result] von Ungern-Sternberg BS, Regli A, Frei FJ, Hammer J, Schibler A, Erb TO. The effect of caudal block on functional residual capacity and ventilation homogeneity in healthy children. Anaesthesia. 2006 Aug;61(8):758-63. doi: 10.1111/j.1365-2044.2006.04720.x. PMID 16867088
- [Result] Singer F, Houltz B, Latzin P, Robinson P, Gustafsson P. A realistic validation study of a new nitrogen multiple-breath washout system. PLoS One. 2012;7(4):e36083. doi: 10.1371/journal.pone.0036083. Epub 2012 Apr 27. PMID 22558338
- [Result] Robinson PD, Goldman MD, Gustafsson PM. Inert gas washout: theoretical background and clinical utility in respiratory disease. Respiration. 2009;78(3):339-55. doi: 10.1159/000225373. Epub 2009 Jun 12. PMID 19521061
- [Derived] Sudy R, Dereu D, Lin N, Pichon I, Petak F, Habre W, Albu G. Respiratory effects of pressure support ventilation in spontaneously breathing patients under anaesthesia: Randomised controlled trial. Acta Anaesthesiol Scand. 2024 Mar;68(3):311-320. doi: 10.1111/aas.14350. Epub 2023 Nov 3. PMID 37923301